CLINICAL TRIAL: NCT00966641
Title: "A Single-Dose Crossover Oral Bioequivalence Study of PL 3100 and Naproxen in Healthy Adult Volunteers in the Fasted State"
Brief Title: Oral Bioequivalence Study of PL 3100 and Naproxen in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL-NAP-001; NIH Grant 1R44AR056529-01
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PL 3100 (Experimental): Active experimental drug
  Interventions: Drug: PL 3100
- Naproxen (Active Comparator): Active comparator
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Single orally administered dose of 500 mg naproxen
  Arms: Naproxen
Drug: PL 3100 — Single orally administered dose of PL 3100 (500 mg naproxen)
  Other Names: Naproxen-PC
  Arms: PL 3100

SUMMARY:
The purpose of this study is to determine the single-dose pharmacokinetics of the investigational drug PL 3100 following oral administration to healthy volunteers and to compare the pharmacokinetic profiles of PL 3100 and naproxen at a prescription dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, inclusive.
* Subject has a Body Mass Index (BMI) between 20 and 32, inclusive.
* Normal physical examination as determined by the Investigator.
* Normal clinical laboratory test results or clinically insignificant results as determined by the Investigator during the screening visit.
* If female and of child-bearing potential, the subject must have a negative pregnancy test and is not nursing.
* If female and of child-bearing potential, the subject must agree to use adequate birth control for the duration of the study.

Exclusion Criteria:

* Subject has a history of chronic alcohol consumption or abuse of narcotics or alcohol.
* Subject has had an acute illness within 5 days of study medication administration.
* Subject is currently participating, or has participated within 30 days prior to study entry, in an investigational drug study.
* Subject has hypersensitivity or contraindications to naproxen, ibuprofen, or other NSAID.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Upendra K. Marathi, PhD, Principal Investigator — PLx Pharma Inc.
Locations (1):
- Houston Institute for Clinical Research, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PL3100 First, Then Naproxen: First Intervention Period:
  PL3100 Capsules: Single orally administered dose of PL 3100 (500 mg naproxen)
  (after 7-14 day washout period)
  Second Intervention Period:
  Naproxen: Single orally administered dose of 500 mg naproxen
- Naproxen First, Then PL3100: First Intervention Period:
  Naproxen: Single orally administered dose of 500 mg naproxen
  (after 7-14 day washout period)
  Second Intervention Period:
  PL3100 Capsules: Single orally administered dose of PL 3100 (500 mg naproxen)
Period: First Intervention
Arm/Group | PL3100 First, Then Naproxen | Naproxen First, Then PL3100
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | PL3100 First, Then Naproxen | Naproxen First, Then PL3100
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants who were enrolled in the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Plasma Naproxen From 0 to t
Description: Blood samples for evaluation of PK variables were collected over a 48-hour period after drug administration.
Time Frame: 30 minutes prior to administration; 30, 60, and 90 minutes post drug administration; and 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, and 48 hours post drug administration.
Population: Pharmacokinetic (PK) Evaluable Population consists of the 28 subjects who completed the study with no protocol deviations.
Measure: Mean (Full Range); unit: min×μg/mL
Arm/Group | PL 3100 | Naproxen
Number analyzed (Participants) | 28 | 28
min×μg/mL | 67763.0 [38832.6 to 100019.6] | 69427.9 [39529.0 to 93963.1]

ADVERSE EVENTS:
Arm/Group | PL 3100 | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 1/34 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL 3100 (N=34) | Naproxen (N=34)
Elevated Partial Thromboplastin Time (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard Confidentiality Agreement